CLINICAL TRIAL: NCT05629364
Title: A Multi-Centre, Randomised, Controlled, Masked Phase 2 Study of the Safety and Efficacy of KIO-101 Ophthalmic Solution, Versus Vehicle Control in the Treatment of Dry Eye Disease in Patients With Autoimmune Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely but potentially will resume
Sponsor: Kiora Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KIO-101-2201
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.15% KIO-101 (Experimental): .15% KIO-101 eyedrops
  Interventions: Drug: KIO-101
- 0.3% KIO-101 (Experimental): 0.3% KIO-101 eyedrops
  Interventions: Drug: KIO-101
- Vehicle (Placebo Comparator): Vehicle eyedrops
  Interventions: Drug: KIO-101

INTERVENTIONS:
Drug: KIO-101 — Randomized, Controlled
  Other Names: DHODH inhibitor

SUMMARY:
A Multi-Centre, Randomised, Controlled, Masked Phase 2 Study of the Safety and Efficacy of KIO-101 Ophthalmic Solution, versus Vehicle Control in the treatment of Dry Eye Disease in Patients with Autoimmune Disease

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of autoimmune disease (psoriatic arthritis, Systemic Lupus Erythematosus (SLE), or fibromyalgia) ≤ 10 years
* Have an Ocular Discomfort Score (ODS) score of ≥3 at Screening
* Have an average VAS score ≥ 50 at Screening; and ≥ 40 at Baseline, Visit 2/Day 1
* Schirmer's 1 test >1 but < 10 mm at Screening.
* National Eye Institute (NEI) corneal fluorescein staining score of ≥ 4 at Screening (Day 14) provided that the total NEI score did not change > ± 2 grades from Screening (Day -14) to Baseline (Day 1) visits, as confirmed by the investigator
* Have a Best Spectacle Corrected Visual Accuity (BSCVA) score of 20/200 (+1.0 LogMAR) or better in both eyes at both the Screening and Baseline visits
* Have a conjunctival hyperaemia score of Grade 2 or more on the Efron Scale in both eyes

Exclusion Criteria:

* Have a history or presence of any ocular disorder or condition (other than dry eye disease (DED)) in either eye that would, in the opinion of the investigator, likely interfere with the interpretation of the study results or subject safety
* Have an autoimmune based vasculitis
* Have a history of RA > 10 years.
* Have a Schirmer's 1 test score of 0 to 1mm at Screening
* Have had a corneal transplant in either or both eyes
* Have had puncta or intracanalicular plug present in either eyelid within 1 year prior to the Screening Visit or anticipated plug insertion or occlusion at any time during the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer's 1 test | 12 weeks
  Change from Baseline to Week 12 for Schirmer's 1 test

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hinds, Principal Investigator — Ophthalmic Trials Australia
Locations (1):
- Ophthalmic Trials Australia, Teneriffe, Queensland, Australia